CLINICAL TRIAL: NCT03556111
Title: Patient Satisfaction and Bone Gain Following Autogenous Particulate Sticky Bone Preparation With Xenograft Versus Without Xenograft for Grafting of Maxillary Anterior Knife-edge Ridge in Partially Edentulous Patients for Implant Placement
Brief Title: Patient Satisfaction and Bone Gain Following Autogenous Particulate Sticky Bone Preparation With Xenograft Versus Without Xenograft for Grafting of Maxillary Anterior Knife Edge Ridge in Partially Edentulous Patients for Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mattar, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sticky bone augmentation
Record Dates: First submitted 2018-04-03; First posted 2018-06-14 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Alveolar Bone Loss; Bone Graft; Complications
Keywords: implant , sticky bone
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anterior knife-edge maxilla graft (Without Xenograft Usage) (Experimental): The intervention will be a Sticky bone augmentation of defect. It is prepared using particulate autologous graft only along with fibrin glue and growth factors obtained from the patients' blood.
  The sample is withdrawn and placed in plastic tubes which are spun twice in a centrifuge at a certain speed and time. The first spin to obtain the fibrin glue and the second to obtain the growth factors. The mixture is added to the harvested autogenous bone to form a semi-solid bone graft that is easily manipulated in the recipient site.
  Interventions: Procedure: Sticky bone augmentation
- anterior knife edge maxilla graft (With Xenograft Usage) (Experimental): The intervention will be the sticky bone augmentation of the defect using both particulate autogenous and xenograft bovine bone.
  The bone will be harvested from the donor, coupled with the bovine bone, the growth factors and the fibrin glue that is obtained from the patient's own blood sample.
  The venous blood sample is placed in plastic tubes to be centrifuged at a certain speed and time to obtain the fibrin glue and growth factors.
  The mixture is prepared until the bone is sticky and ready to be placed in the recipient defective maxilla
  Interventions: Procedure: Sticky bone augmentation

INTERVENTIONS:
Procedure: Sticky bone augmentation — 1. Autogenous sticky bone augmentation for the first group
  2. Autogenous sticky bone preparation with xenograft usage
  3. After 5-month of bone grafting; esthetic implant placement

SUMMARY:
The aim is to evaluate the value and efficiency of sticky bone in the augmentation of alveolar ridge deficiency when being used with or without xenogenic bone graft for esthetic implant placement.

DETAILED DESCRIPTION:
Modern Dentistry aims to restore what is missing, no matter what the difficulty is. As many patients have lost their teeth to a number of factors, either trauma or disease or lack of care. Now the individuals are seeking to restore the function and esthetics. The more the number of teeth is missing along with ridge deficiencies can present serious challenges to the clinician.

Implant supported prosthesis is an attractive option for restoring edentulous or partially edentulous patients. However, extensive loss of the alveolar bone is a complex problem that faces many surgeons. This era has witnessed numerous trials and research for bone augmentation for the defective alveolar ridge. The goal is to create sufficient space for endosseous implant placement in a knife edge ridge.

Alveolar bone resorption occurs in either a horizontal or vertical direction. It can also be composite. There are 3 classes of bone-grafting materials based upon the mode of action. Autogenous bone is an organic material and forms bone by osteogenesis, osteoinduction, and osteoconduction.

Allografts such as demineralized freeze-dried bone are osteoinductive and osteoconductive and may be cortical and/or trabecular in nature.

Alloplasts such as hydroxyapatite and tricalcium phosphate may be synthetic or natural, vary in size, and are only osteoconductive. They can be divided into three types based upon the porosity of the product and include dense, macroporous, and microporous materials. In addition, alloplastic materials may be crystalline or amorphous. These materials have different properties and therefore indications.

Previous studies have shown that although the autogenous bone is considered as the Gold Standard of bone grafting for its osteogenic potential, many drawbacks exist which limits its application. For instance, donor site morbidity is of concern. Bone harvesting procedures may put adjacent anatomical structures at a risk of damage. During chin bone harvesting, the mental nerve may be pulled under undue traction and the incisive nerve become interrupted when the harvesting depth is inordinate. Ramus bone harvesting can damage the inferior alveolar nerve. In addition, some patients may be reluctant to the harvesting procedures, especially when extra-oral donor sites are concerned. General anesthesia is mandatory for such operations.

Recent research studies have looked into modifying the surgical techniques in order to regain the space for an implant along with finding satisfying esthetic outcomes. The literature shows the positive use of ridge splitting technique and alveolar distractors, with or without the aid of xenograft material and/or alloplastic material.

Starting from the early 2000s, a new drift of guided bone regeneration research blew by. Platelet concentrates (PC); platelet-rich plasma (PRP) and platelet-rich fibrin (PRF)] were used for surgical procedures in medical and dental fields, particularly in Oral and Maxillofacial surgery, plastic surgery and sports medicine.

They were utilized to accelerate healing of bone graft over the bony defects, many techniques utilizing platelet and ﬁbrinogen concentrations have been introduced in the literature. Platelet is known to contain high quantities of growth factors, such as transforming growth 4 . Factors ß-1 (TGFß-1), platelet-derived growth factor (PDGF), epithelial growth factor (EGF), insulin growth factor-I (IFG-I) and vascular endothelial growth factors (VEGF), which stimulates cell proliferation and upregulates angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* - Alveolar bone width 3mm or less in anterior maxillary knife edge ridge as evaluated preoperatively on the CBCT
* Both sexes.
* Good oral hygiene.
* Age between 18 and 48 years. Highly motivated patients

Exclusion Criteria:

* - Patient with Bad oral hygiene
* Post-menopausal females with osteoporosis
* Patient with uncontrolled systemic disease For instance: uncontrolled Diabetes Mellitus

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 8 months after bone graft placement
  Patient satisfaction with the bone gain and the prosthetic implant placement

SECONDARY OUTCOMES:
bone width gain | 5 month after bone graft placement
  measured in mm
Successful implant placement | 5 months after bone graft placement
  it will be measured using OsstellISQ

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry , Cairo University., Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR